CLINICAL TRIAL: NCT04770597
Title: Monitors to Improve Indoor Carbon Dioxide (CO2) Concentrations in the Hospital: a Randomized, Sham-controlled, Open Label Trial
Brief Title: Monitors to Improve Indoor Carbon Dioxide (CO2) Concentrations in the Hospital
Acronym: MICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imelda Hospital, Bonheiden (Other)
Responsible Party: Principal Investigator, Michaël R Laurent, MD PhD, Principal Investigator, Imelda Hospital, Bonheiden
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20210209
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Healthcare Associated Infection
Keywords: Indoor air quality; Carbon dioxide; Ventilation
MeSH Terms: conditions — Cross Infection; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Each sensor will be randomized to Sham-Intervention or Intervention-Sham cross-over. Additionally, each sensor will measure CO2 during a baseline and post-intervention phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): CO2 values on sensor visible to staff
  Interventions: Device: Aranet4 Home CO2 monitor
- Sham control (Sham Comparator): CO2 values on sensor not visible to staff
  Interventions: Device: Aranet4 Home CO2 monitor

INTERVENTIONS:
Device: Aranet4 Home CO2 monitor — The sensor is placed in the room at a height between 1 and 2 meters and not near the window or door.

SUMMARY:
Ventilation with fresh outdoor air has recently gained considerable attention as a means to reduce the potential risk of indoor aerosol transmission of respiratory pathogens such as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus causing coronavirus disease 2019 (COVID-19). Commercial carbon dioxide (CO2) monitors are increasingly used in schools, long-term care facilities, offices and public buildings to monitor indoor ventilation. However, no formal evidence is available to support the effectiveness of feedback from CO2 monitoring devices. Moreover, modern hospitals have superior indoor air quality control systems.

The aim of this prospective pilot randomized controlled trial (RCT) is to evaluate whether CO2 monitoring devices would be useful as a means to further maintain lower indoor CO2 concentrations in hospitals.

DETAILED DESCRIPTION:
In this pilot, randomized, sham-controlled open-label RCT, hospital rooms will be fitted with Aranet4 Home CO2 sensors.

Each device will continuously measure indoor CO2 concentrations at 1-minute intervals during 4 time periods:

1. Baseline: staff blinded to CO2 levels displayed on sensor

2-3. Sham/Intervention period: sensors on the same ward will be randomized to placebo (sensor not showing CO2 levels to staff) or Intervention (sensor displaying CO2 levels to staff) in a cross-over design

4. Post-intervention phase (3 weeks post-intervention): staff blinded to CO2 levels

Each measurement period will consist of 7 days with no washout period.

Our primary hypothesis is that CO2 sensors will record less time (minutes) with elevated CO2 levels during the intervention period, compared to the Sham periods. However, carry-over effects will be investigated by comparing the Intervention periods to the Baseline and Post-intervention phases.

Note [February 27, 2021]: due to technical problems with the Aranet4 device Bluetooth connection, outcome data will be analyzed according to measurement data at 2-5 minute intervals (measurements can be made every minute, but data cannot be downloaded with the current version of the app due to technical problems).

ELIGIBILITY:
Inclusion Criteria:

* Double-bed hospital rooms

Exclusion Criteria:

* Unoccupied rooms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — When applicable, patients stay in double-bed rooms based on gender.
Enrollment: 12 (Actual)
Dates: Start 2021-02-21 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
Time >800 ppm CO2 | 7 days/time period (pre-, active/sham and post-intervention)
  Time/day (in minutes/24h) measuring >800 ppm CO2

SECONDARY OUTCOMES:
Time >1000 ppm CO2 | 7 days/time period (pre-, active/sham and post-intervention)
  Time/day (in minutes/24h) measuring >1000 ppm CO2
Time >1400 ppm CO2 | 7 days/time period (pre-, active/sham and post-intervention)
  Time/day (in minutes/24h) measuring >1400 ppm CO2
Daily peak CO2 concentration [in ppm] | 7 days/time period (pre-, active/sham and post-intervention)
  Daily peak CO2 concentration [in ppm]

OTHER OUTCOMES:
Staff-rated feasibility on a 10-point Likert scale [0-10, with 10 indicating better outcome] | 7 days
  How feasible is it to use CO2 sensors to monitor indoor air quality in hospital? Anonymous online survey during the post-intervention phase
Staff-rated preference on a 10-point Likert scale [0-10, with 10 indicating better outcome] | 7 days
  Would you prefer to use CO2 sensors to monitor indoor air quality in hospital in the future? Anonymous online survey during the post-intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Michaël R Laurent, MD PhD, Principal Investigator — Geriatrics Department, Imelda Hospital Bonheiden
Locations (1):
- Imelda Hospital, Bonheiden, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The full set of sensor data will be made available to established investigators upon simple request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available upon fulltext print publication in a peer-reviewed journal, for a duration of at least 10 years.
Access Criteria: Simple e-mail request to the corresponding author by an established scientific investigator

REFERENCES:
- [Derived] Laurent MR, Frans J. Monitors to improve indoor air carbon dioxide concentrations in the hospital: A randomized crossover trial. Sci Total Environ. 2022 Feb 1;806(Pt 3):151349. doi: 10.1016/j.scitotenv.2021.151349. Epub 2021 Oct 30. PMID 34728206